CLINICAL TRIAL: NCT07212894
Title: The Effect of DemensiaKITA Mobile Health Application Intervention on Knowledge, Attitude, Practice (KAP) and Burden Level of Dementia Caregivers in Kuala Lumpur and Selangor, Malaysia: Protocol for a Non-Randomized Controlled Trial
Brief Title: DemensiaKITA Mobile Health App to Improve Knowledge, Attitude, Practice and Reduce Burden Among Dementia Caregivers in Malaysia
Acronym: DemensiaKITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Nurulizzah binti Mahfar, Doctor, Universiti Teknologi Mara
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UiTM-DemCareKAP-2025; UiTM-FERC/25/600-TNCPI (5/1/6) (Other: Universiti Teknologi MARA (UiTM))
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Dementia
Keywords: Dementia; Informal Caregivers; Mobile health application; Knowledge Attitude Practice; Burden level; Malaysia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model with two groups. Dementia caregivers in the intervention group will receive access to the DemensiaKITA mobile health application, which provides structured educational modules, caregiving practice tips, and self-monitoring tools. Caregivers in the control group will continue with usual care and standard support resources available in the community. Outcomes will be assessed in both groups at baseline and after the intervention period to evaluate differences in knowledge, attitude, practice, and caregiver burden.
Who Masked: Participant
Masking Description: This is a non-randomized, single-blinded study. Participants are blinded to their group assignment (intervention or control). Care providers and investigators are aware of the allocation, but participants are not informed which group they belong to in order to reduce bias in outcome reporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Intervention): DemensiaKITA mHealth app (Experimental): Arm 1: DemensiaKITA Mobile Health App
  Arm Description:
  Participants in this arm will receive access to the DemensiaKITA mobile health application. The app delivers structured dementia-related education, strategies to improve caregiver knowledge, positive attitude reinforcement, and practical caregiving tips. It also provides self-monitoring features to support caregiver well-being. Participants will be encouraged to use the application regularly throughout the study period.
  Interventions: Other: DemensiaKITA mobile health application
- Arm 2 (Control): Usual care (Experimental): Arm 2: Usual Care
  Arm Description:
  Participants in this arm will continue with their usual caregiving practices and community resources. They will not have access to the DemensiaKITA mobile health application during the study period. This group serves as the comparator to evaluate the effectiveness of the intervention.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: DemensiaKITA mobile health application — A mobile health application developed to support dementia caregivers. It provides structured educational modules, attitude-shaping content, and practical caregiving tips, along with self-monitoring features to reduce caregiver stress and burden. Participants in the intervention group will use the app regularly during the study period.
  Arms: Arm 1 (Intervention): DemensiaKITA mHealth app
Other: Usual Care — Participants assigned to the control group will continue with usual caregiving practices and community-based resources available to dementia caregivers. They will not be given access to the DemensiaKITA mobile health application during the study period. This group provides a comparator for evaluating the added benefit of th
  Arms: Arm 2 (Control): Usual care

SUMMARY:
Dementia is a growing health concern in Malaysia and places a heavy burden on family members who act as caregivers. Many caregivers struggle with limited knowledge, negative attitudes, and challenges in daily caregiving practices. These issues increase caregiver stress and reduce the quality of care for people living with dementia.

The DemensiaKITA mobile health application was developed to support caregivers by providing educational content, self-help tools, and practical guidance. This study will evaluate whether using the DemensiaKITA app can improve caregivers' knowledge, attitudes, and caregiving practices (KAP), as well as reduce caregiver burden.

This is a non-randomized controlled trial involving dementia caregivers in Kuala Lumpur and Selangor. Participants in the intervention group will use the DemensiaKITA mobile app for a set period, while the control group will continue with usual support. Outcomes will be measured before and after the intervention using validated questionnaires.

The results of this study will provide evidence on the effectiveness of a locally developed mobile health application in supporting dementia caregivers in Malaysia. If successful, this digital approach may be scaled up to improve caregiver support and dementia care in other settings.

DETAILED DESCRIPTION:
The rising prevalence of dementia in Malaysia has increased the need for caregiver support strategies. Informal caregivers often face knowledge gaps, negative perceptions, and poor caregiving skills, collectively referred to as Knowledge, Attitude, and Practice (KAP) challenges. Additionally, caregiver burden is a well-documented consequence of long-term dementia care, leading to stress and reduced quality of life.

The DemensiaKITA mobile health application was designed to provide accessible, structured, and culturally relevant caregiver education. Its features include dementia-related knowledge modules, attitude-shaping messages to encourage empathy and positive caregiving, and practice tips for daily care. It also offers self-monitoring tools to track caregiving challenges and support caregiver well-being.

This non-randomized controlled trial will recruit dementia caregivers from Kuala Lumpur and Selangor. Participants will be allocated into intervention and control groups. The intervention group will use the DemensiaKITA app for a defined duration, while the control group will receive usual care and information. Pre- and post-intervention data will be collected using validated instruments such as the Dementia Knowledge Assessment Tool (DKAT-2), caregiver attitude and practice scales, and the Zarit Burden Interview (ZBI).

Primary outcomes include improvements in KAP scores, while secondary outcomes include reductions in caregiver burden. The study findings will inform the potential integration of mobile health applications into community-based dementia support programs in Malaysia and similar low- and middle-income country settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Primary informal caregiver of a person living with dementia (family member or household member)
* Able to read and understand Malay
* Owns a smartphone and is able to use mobile applications
* Provides informed consent to participate

Exclusion Criteria:

* Professional/paid caregivers (e.g., nurses, domestic helpers hired solely for caregiving)
* Caregivers of patients with conditions other than dementia
* Individuals with severe cognitive or psychiatric illness that limits their ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 451 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dementia Caregivers' Knowledge, Attitude, and Practice (KAP) Scores | Baseline, 1 month and 3 months after intervention start
  Caregiver knowledge, attitude, and practice will be assessed using validated instruments, including the Dementia Knowledge Assessment Tool (DKAT-2) and caregiver attitude and practice scales. The primary outcome is the change in KAP scores between baseline and post-intervention, comparing the intervention (DemensiaKITA app) and control (usual care) groups. Higher scores indicate better knowledge, more positive attitudes, and improved caregiving practices.

SECONDARY OUTCOMES:
Change in Caregiver Burden Scores | Baseline, 1 month and 3 months after intervention start
  Caregiver burden will be measured using the Zarit Burden Interview (ZBI), a validated questionnaire assessing the level of stress, emotional strain, and impact of caregiving responsibilities. The outcome is the change in ZBI scores between baseline and post-intervention. Lower scores indicate reduced caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Nurulizzah Mahfar, Principal Investigator — Universiti Teknologi MARA Sg Buloh Campus
Locations (1):
- Universiti Teknologi MARA, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data (IPD) due to ethical considerations and data protection regulations in Malaysia. The data involve informal caregivers of persons living with dementia, a population considered vulnerable. Sharing de-identified datasets may still pose a risk of re-identification, especially given the relatively small sample size and localized recruitment sites. Instead, study findings will be disseminated through peer-reviewed publications, conference presentations, and summary results reported on ClinicalTrials.gov, ensuring transparency while protecting participant confidentiality.